CLINICAL TRIAL: NCT06300736
Title: HEPIC Study : Design of a Predictive Score for Contamination of Pediatric Blood Cultures
Brief Title: Design of a Predictive Score for Contamination of Pediatric Blood Cultures
Acronym: HEPIC
Status: Active, not recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GIROUX Nathan, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2023PI247
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Bacteremia
Keywords: Blood culture contamination; Predictive score
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The contamination rate for blood cultures is high in pediatrics, due to different sampling techniques and the difficulty of sampling small-weight children, thus favoring contamination of the devices at the time of sampling. It is also more difficult to distinguish contamination from true bacteremia in children at an early stage, notably due to the limited number of vials that can be taken at any one time.

On a daily basis, clinicians are faced with the choice of whether or not to initiate probabilistic antibiotic therapy when faced with the result of a positive blood culture, particularly when identification is not yet available, but only direct examination.

Contamination has major consequences for patient management. Studies in adults have shown that contamination increases hospital length of stay by 4 to 5 days, laboratory costs by +20% and recourse to intravenous antibiotic therapy by +39%. In children, studies came to the same conclusion, with greater prescription of antibiotics, particularly intravenous antibiotics, in patients with contaminated blood cultures than in patients with sterile blood cultures. It also showed that 26% of patients with contaminated blood cultures were initially hospitalized because of the positivity of this test.

The aim of this research is to determine the factors associated with contamination, in order to create a predictive score that would help clinicians in their decision-making when receiving the blood culture result as "positive".

ELIGIBILITY:
Inclusion Criteria:

* Having a blood culture in children's hospital in Nancy
* Under 18 years old
* in emergency department, medical department, intensive care unit or surgical department

Exclusion Criteria:

* immunodepression
* post mortem blood culture
* blood culture in onco-haematology department

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Immunocompetent children hospitalized in a tertiary children hospital with blood culture
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Blood culture diagnosis | 2 years
  Contamination or bacteriemia

SECONDARY OUTCOMES:
Score performance | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nathan GIROUX, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU Nancy, Nancy, France